CLINICAL TRIAL: NCT06634199
Title: Study of Antitumor Immune Response Generated After Concurrent Chemo-radiotherapy (cCRT) and IO Treatment in Non-resectable Stage IIIA/B and IIIC NSCLC Patients Treated in Real World.
Brief Title: Study of Antitumor Immune Response After cCRT and IO Treatment in Non-resectable III Stage NSCLC Patients
Acronym: SIENNA
Status: Recruiting | Type: Observational
Sponsor: Fundación GECP (Other)
Responsible Party: Sponsor
Other Study IDs: GECP 23/04_SIENNA
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer Stage III; PDL1 Gene Mutation
Keywords: Lung Cancer; Chemo radiotherapy; ctDNA; Inmunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — durvalumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Archival tumor samples Routine Blood samples extraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Study Group: Real world non-small cell lung cancer (NSCLC) stage IIIA/B and IIIC; PD-L1>1%; non-resectable patients in treatment with IO after concurrent chemo-radiotherapy without progression.
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — Chemo-radiotherapy + Durvalumab for non-resectable stage III NSCLC patients according to clinical practice of each participant hospital
  Other Names: Imfinzi

SUMMARY:
Observational, multicenter, one-arm, non-comparative study. Data will be recorded in a retrospectively manner. The study will be based on secondary data collected from patient clinical chart completed by the doctor during routine visits. The primary objective is describe the antitumor immune response generated in the context of IO (immunotherapy) treatment after cCRT in patients with unresectable NSCLC treated in real world.

DETAILED DESCRIPTION:
The study is based on the collection of blood samples and tumor sample analysis, in real world NSCLC stage IIIA/B and IIIC; PD-L1>1%; non-resectable patients on treatment with IO after cCRT without progression. The patients participating in this study will not receive treatment in relation to the study, no drugs will be provided. Patients will be treated as per standard clinical practice. All data collected for this study will be collected retrospectively from patient clinical chart. Only secondary data collected will be analyzed together will samples analysis information.The duration of the study is expected to be 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically- or cytologically- documented NSCLC who present unresectable stage IIIA-IIIB-IIIC disease, according to 8th version of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology).
* ECOG 0-1.
* PDL1>1%.
* Age ≥ 18 years at time of study
* Patients without progression after cCRT, that are going to receive IO treatment (Durvalumab) for 12 months as subsequent treatment as per standard clinical practice
* Patient capable of proper therapeutic compliance and accessible for correct follow-up.
* Patients must have signed, dated and IRB/EC-approved written informed consent form in accordance with regulatory and institutional guidelines.

Exclusion Criteria:

* Patients who refuse to sign and date an IRB/IEC-approved written informed consent form.
* No possibility of venipuncture
* Any medical, mental, or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or understand the patient information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Real world non-small cell lung cancer (NSCLC) stage IIIA/B and IIIC; PD-L1>1%; non-resectable patients in treatment with IO after concurrent chemo-radiotherapy without progression.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2027-11-04 (Estimated); Study Completion 2027-11-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | To evaluate the Overall Survival at 12, 18, 24 and 36 months
  Defined from the date of diagnosis to death from any cause. Patients alive at the end of follow-up or lost to follow-up are censored at the last contact time. The probability of remaining free of events at specific timepoints
Progression-free survival (PFS) | To evaluate the Progression-free survival at 12, 18, 24 and 36 months
  Defined from the diagnosis date to the date of investigator-determined disease relapse or death, whichever occurs first. The probability of remaining free of events at specific timepoints

SECONDARY OUTCOMES:
Association between ctDNA clearance (no detection of ctDNA) after IO treatment and Progression free survival (PFS) or Overall survival (OS). | From date of end of treatment until the date of last follow up, assessed up to 36 months
  Association between the baseline ctDNA and ctDNA clearance with each one of the OS or PFS

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Provencio, MD, Study Chair — Fundación GECP President
Locations (22):
- Spain (22):
  - Complejo Hospitalario Universitario Del Ferrol, Ferrol, A Coruña
  - Hospital General Universitario de Alicante, Alicante, Alicante
  - ICO Badalona, Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari Vall d' Hebron, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital De Basurto, Bilbao, Bilbao
  - Hospital General Universitario de Ciudad Real, Ciudad Real, Ciudad Real
  - ICO Girona, Hospital Josep Trueta, Girona, Girona
  - Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Hospital Universitari de Gran Canària Doctor Negrín, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Lucus Augusti, Lugo, Lugo
  - Hospital Universitario De La Princesa, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario Central De Asturias, Oviedo, Oviedo
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife, Santa Cruz de Tenerife
  - Hospital Virgen del Rocio, Seville, Sevilla
  - Hospital Universitario Y Politécnico La Fe, Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid, Valladolid
  - Complexo Hospitalario Universitario De Vigo, Vigo, Vigo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org